CLINICAL TRIAL: NCT05002751
Title: Quantifying Radiation Induced Vaginal Stenosis for the Development of a Novel Dilator Device
Brief Title: Quantifying Radiation Induced Vaginal Stenosis
Acronym: QRIVS
Status: Recruiting | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jyoti Mayadev, MD, Associate Professor, University of California, San Diego
Other Study IDs: QRIVS-001; PAR 20-292 (Other: National Istitutes of Healh (NIH)); PAR 20-292 (Other: National Cancer Institute (NCI))
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Vaginal Stricture; Vaginal Stenosis
Keywords: Vaginal Stenosis; Vaginal Stricture; Radiotherapy Side Effect; Brachytherapy Side Effect
MeSH Terms: conditions — Radiation Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: 1. Patients with histologically confirmed newly diagnosed advanced cervical cancer (squamous cell carcinoma, adenocarcinoma, and adenosquamous cell carcinoma): FIGO 2009 clinical stages IB2/IIA with positive para-aortic nodes, or FIGO 2009 clinical stages IIB/IIIB/IVA with positive pelvic or para-aortic lymph nodes (PALN). Pelvic or PALN nodal status confirmed by PET/CT scan or fine needle biopsy or extra peritoneal biopsy or laparoscopic biopsy. The PALN must be inferior to the T12/L1 interspace.
  Interventions: Other: UCSD Vaginal Dilator Questionnaire; Other: EORTC Sexual Health Questionnaire

INTERVENTIONS:
Other: UCSD Vaginal Dilator Questionnaire — 14 question survey
Other: EORTC Sexual Health Questionnaire — 22 question survey

SUMMARY:
Radiation (RT) affects the vagina by narrowing, tightening and scarring, termed vaginal stenosis (VS). VS occurs in up to 88% of patients treated with radiation for cervical cancer. VS is not well characterized in measurements. There is a lack of understanding of how short and tight the vagina becomes after RT. This study will use specific measurements of the vagina during the routine physician physical exam after RT in the follow up periods: after RT, 3 months, 6 months, and 12 months using a plastic commercial dilator set and length and width measurements.

In addition, the study use a validated sexual health survey and a specific survey on vaginal dilation preferences to help stop VS after RT.

DETAILED DESCRIPTION:
This single-arm pilot will enroll 12 subjects scheduled to receive radiotherapy or brachytherapy for gynecological cancers. The study will collect data from CT images, physical measurements, patient reported outcomes to develop a quantifiable generalizable metric for determining the severity of radiotherapy/brachytherapy induced vaginal stenosis.

The data will be used to inform the development of a novel personalized device for the treatment of vaginal stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed newly diagnosed advanced cervical cancer (squamous cell carcinoma, adenocarcinoma, and adenosquamous cell carcinoma): FIGO 2009 clinical stages IB2/IIA with positive para-aortic nodes, or FIGO 2009 clinical stages IIB/IIIB/IVA with positive pelvic or para-aortic lymph nodes (PALN). Pelvic or PALN nodal status confirmed by PET/CT scan or fine needle biopsy or extra peritoneal biopsy or laparoscopic biopsy. The PALN must be inferior to the T12/L1 interspace.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix II).
* Patients must have normal organ and marrow function as defined below:

  1. leukocytes ≥2,500/mcL
  2. absolute neutrophil count ≥1,500/mcL
  3. platelets ≥100,000/mcL
  4. hemoglobin ≥8 g/dL (can be transfused with red blood cells pre- study)
  5. total bilirubin ≤1.5 × institutional upper limit of normal (ULN)
  6. AST(SGOT)/ALT(SGPT) ≤3 × ULN
  7. alkaline phosphatase ≤2.5 × ULN
  8. creatinine <1.5 mg/dL INR and aPTT ≤1.5 × ULN (This applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation, such as low-molecular-weight heparin or warfarin, should be on a stable dose.)
* Age is > 18 years.
* Patient does not have a known allergy to cisplatin or compounds of similar biologic composition.
* Ability to understand and the willingness to sign a written informed consent document.
* Patients positive for human immunodeficiency virus (HIV) are allowed on study, but HIV-positive patients must have:
* A stable regimen of highly active anti-retroviral therapy (HAART)
* No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
* A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard PCR-based tests.

Exclusion Criteria:

* Patients who have received prior radiation therapy to the pelvis or abdominal cavity, PALN radiation, or previous therapy of any kind for this malignancy or pelvic, PALN, or abdominal radiation for any prior malignancy.
* Patients with PALN nodal metastasis above the T12/L1 interspace.
* Patients who had a radical hysterectomy with positive PALNs are not eligible.
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation.
* Patients previously treated with systemic anticancer therapy (e.g., chemotherapy, targeted therapy, immunotherapy) within 3 years prior to entering the study.
* Patients diagnosed on imaging or biopsy with a synchronous primary malignancy (with the exception of DCIS of the breast, or early stage basal cell carcinoma of the skin)

  a. transcription mediated amplification (TMA) or branched DNA testing.
* History or risk of autoimmune disease, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female subjects over 18 years old, scheduled to receive radiotherapy and/or brachytherapy for the treatment of gynecological cancers.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2022-10-06 (Actual); Primary Completion 2026-04-05 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Quantify radiation induced vaginal stenosis | 1.5 years
  acquire and integrate imaging and direct patient vaginal diameter measurements to characterize VS for the computer and benchtop models
Acquire Patients' Treatment Concerns and Preferences | 1.5 years
  Using a series of sexual and vaginal health questionnaires presenting an array of scaled (quantified) options we will determine patients' perceived flaws about current treatment and their preferences, and integrate them with the VS measurement results of Aim1 to guide modification and optimization of our soft balloon VS treatment system
Optimize and Validate Vaginal Stenosis Treatment System | 1 year
  Incorporating the multimodal vaginal stenosis measurements and patient preferences acquired in Aim 1, we will use computer modelling based on known vaginal wall properties to simulate and predict the long-term outcomes of balloon-driven, graded vaginal expansion to counteract VS. Benchtop experimentation will utilize an inflatable balloon-type device and 3D printed biomimetic stenosed vaginal phantoms to test the proposed treatment effect over various time periods emulating different stages of fibrotic stenosis. To directly test our working hypothesis results acquired from modeling will be compared statistically to benchtop data.

CONTACTS AND LOCATIONS:
Overall Officials: Jyoti Mayadev, MD, Principal Investigator — University of California, San Diego Moores Cancer Center
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No